CLINICAL TRIAL: NCT02794896
Title: Hypnotic Depth Reduces Lymphocyte Proliferation to Natural Killer Cells, B-cells, Memory T-cells, Depresses Intracellular Oxidative Burst and Changes Protein Expression Pattern of Monocytes
Brief Title: Anesthetic Depth Effects Upon Immune Competent Cells
Acronym: BIS-MA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Thomas Frietsch, Associate Professor of the Dept. of Anesthesiology and Critical Care Medicine, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Anesthetic depth-MA
Record Dates: First submitted 2016-05-12; First posted 2016-06-09 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Immunotoxicity; Anesthesia; Inert Gas Narcosis
MeSH Terms: conditions — Inert Gas Narcosis | interventions — Propofol; Fentanyl; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep Anesthesia (Experimental): Standard anesthesia with fentanyl, propofol for shoulder surgery together with a interscalene plexus block was performed. The anesthesiologist only was informed about the group allocation by the study director and tried to control best for maintenance on target anesthesia level BIS 45 (group 1, deep anesthesia). Anesthesia depth was measured by BIS monitors (BIS Vista, Aspect) for every minute and the minutes below or equal to a BIS level of 45 were counted.
  Interventions: Drug: High dose propofol, fentanyl and sevoflurane
- Shallow Anesthesia (Experimental): Standard anesthesia with fentanyl, propofol for shoulder surgery together with a inter scalene plexus block was performed. The anesthesiologist only was informed about the group allocation by the study director and tried to control best for maintenance on target anesthesia level BIS ≥ 55 (group 2, shallow anesthesia). Anesthesia depth as measured by BIS monitors (BIS Vista, Aspect) for every minute and the minutes above a BIS level of 45 were counted.
  Interventions: Drug: Low dose propofol, fentanyl and sevoflurane

INTERVENTIONS:
Drug: High dose propofol, fentanyl and sevoflurane — Deep Anesthesia
  Other Names: BIS lower than or equal to 45
  Arms: Deep Anesthesia
Drug: Low dose propofol, fentanyl and sevoflurane — Shallow Anesthesia
  Other Names: BIS above 45
  Arms: Shallow Anesthesia

SUMMARY:
Anesthesia depth affects the proliferation of lymphocytes to NK-cells and memory T-cells effect and the phagocytosis activity of macrophages in healthy patients. ASA 1-3 subjects undergoing extended shoulder surgery under continuous regional anesthesia randomly were assigned to a deep or a shallow anesthesia level (BIS <35 or >55) for more than an hour. Immune response is measured by lymphocyte proliferation as well as neutrophil and monocyte phagocytosis activity.

DETAILED DESCRIPTION:
Blood samples were taken under minimal stress prior to anesthesia induction (T0), recovery (T1) and 12 weeks following hospital discharge (T2) from the respective anesthesia depth level. Bispectral index monitoring (BIS) was performed from the awake state to complete recovery in all subjects.

Hemoglobin concentration, leukocyte and lymphocyte counts were determined by routine automated laboratory techniques. Lymphocyte proliferation was analyzed by SASPA flow cytometry analysis. In brief, 100 µl EDTA blood were stirred with 10 µl FITC and PE marked antibody mixture containing CD3, CD4, CD8, CD 16, CD45, CD28, CD27, CD 56.

Monocyte and neutrophil phagocytosis activity was measured separately in macrophages of fresh heparinized whole blood using flow cytometric test kits.

Proteomics of monocytes was done synchronously.

ELIGIBILITY:
Inclusion Criteria:

* enrolment for longer shoulder surgery
* consent for the standard anesthesia form in combination with the interscalene plexus block
* ASA Status 1-3

Exclusion Criteria:

* sedative premedication
* severe immune deficiency (diabetes, steroid or antihistamine medication, cancer, chemotherapy,
* status post transplantation, drug and alcohol abuse),
* recent surgery (1 month) or blood transfusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Depression of lymphocyte proliferation by CD expression pattern in SASPA-Test as given in a percentage from before anesthesia | 70-90 min
  before and following anesthesia period over 60 min

SECONDARY OUTCOMES:
Reduction of phagocytosis activity as a percentage of base line (prior to anesthesia) | 70-90 min
  before and following anesthesia period over 60 min
Protein expression pattern of monocytes by proteomics analysis and mass spectrometry | 70-90 min
  before and following anesthesia period over 60 min

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frietsch, MD, PhD, Principal Investigator — University of Mannheim
Locations (1):
- University Medicine of Mannheim, Dept. Anesthesiology and Critical Care Medicine, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Yes
per request

REFERENCES:
- [Derived] Nguyen XD, Horn A, Fischer D, Beck G, Spannenberger CC, Gaudilliere B, Horn JL, Thierse HJ, Frietsch T. Suppressive effects of deep balanced anesthesia on cellular immunity and protein expression: a randomized-controlled pilot study. BMC Anesthesiol. 2025 Mar 17;25(1):129. doi: 10.1186/s12871-025-02980-9. PMID 40097954